CLINICAL TRIAL: NCT06457217
Title: Magnetic Resonance Spectroscopic Imaging Evaluation for Understanding Acute Minor Stroke With Large Vessel Occlusion Evolution Study
Brief Title: MRSI Evaluation for Minor Stroke With Large Vessel Occlusion
Acronym: MINORITY
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Li Cao, Professor, Shanghai 6th People's Hospital
Other Study IDs: MRSI20240309(1)
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Magnetic resonance spectroscopic imaging; Clinical Deterioration; Neurotransmitter; Neurometabolite; Metabolic network connectivity
MeSH Terms: conditions — Ischemic Stroke; Clinical Deterioration | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LVO-MIS: Acute minor ischemic stroke induced by large vessel occlusion (LVO-MIS) within 24 hours
  Interventions: Diagnostic Test: Magnetic resonance spectroscopic imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance spectroscopic imaging — High-resolution 3D metabolic imaging was performed using the SPICE 1H-MRSI sequence.

SUMMARY:
The goal of this observational study is to understand acute anterior circulation large artery occluded minor stroke (LVO-MIS) evolution using magnetic resonance spectroscopic imaging evaluation. The main questions it aims to answer are:

1. Neurometabolic predictors of early neurological deterioration and functional outcome;
2. Temporal and spatial dynamic changes of the neurometabolites from the acute stage (within 24 hours), through the subacute stage (5-7 days), to the chronic stage (90 days);
3. Temporal and spatial dynamic changes of the neurotransmitters GABA, glutamate, and glutamine from the acute stage to the chronic stage;
4. Brain regions exhibiting changes in whole-brain metabolic network connectivity.

DETAILED DESCRIPTION:
Minor acute ischemic stroke (AIS) is a common medical condition accounting for more than 50% of AIS. Of the patients with minor AIS, 28.3% are unable to discharge home, and 28.5% cannot walk independently. Although most patients with large vessel occlusion (LVO) strokes and mild symptoms have good clinical outcomes, individuals with early neurological worsening tend to do poorly despite rescue thrombectomy. Therefore, it would be ideal to understand the factors associated with acute neurological deterioration ≥4 NIHSS points among this population to potentially triage higher risk individuals to upfront endovascular therapy.

The main goal of this study was to investigate the spatial and temporal changes of neurometabolite concentrations in patients with acute mild ischemic stroke with large vessel occlusion (LVO-MIS) and to assess the extent to which the combination of all neurometabolite signals measured by 3D-MRSI could discriminate between early neurologic deterioration (END) and non-END patients.

Patients who are older than 18 years of age diagnosed with acute mild ischemic stroke with large vessel occlusion (LVO-MIS) within 24 hours of onset will be enrolled into the study. MRSI will be performed in enrolled stroke patients from the acute stage (within 24 hours), through the subacute stage (5-7 days), to the chronic stage (90 days). Higher resolution 3D MRSI scans were performed using SPICE. The acquisition parameters were as follows: TR = 160 msec, TE = 1.6 msec, spatial resolution = 2.0 × 3.0 × 3.0 mm3, FOV = 240 × 240 × 120 mm3, scan time = 18:35 min.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age ≥ 18 years) patients presenting with symptoms consistent with acute ischemic stroke due to occlusion of the intracranial internal carotid artery and/or M1 or M2 segment of the middle cerebral artery;
2. Patients with mild symptoms at admission (National Institutes of Health Stroke Scale (NIHSS)<6);
3. Baseline multimodal-CT imaging, including NCCT, CTA and CTP, performed at the trial-site hospital;
4. Time from symptom onset or last known normal to enrollment is less than 24 hours;
5. Patient or legal representative willing to comply with protocol requirements and data collection procedures, understand and sign informed consent.

Exclusion Criteria:

1. A pre-incident mRS ≥ 1 point before onset;
2. Previous clear history of cerebral infarction, cerebral hemorrhage, brain tumor and other diseases that affect cerebral metabolism;
3. Intolerance or non-cooperation with magnetic resonance examination;
4. Severe cardiac, hepatic, renal impairment or other systemic serious advanced diseases;
5. Pregnancy or lactation;
6. Life expectancy is less than 3 months;
7. Other conditions that, in the opinion of the investigator, are not suitable for participation in this study or may pose a significant risk to the patient (such as inability to understand and/or comply with study procedures and/or follow-up due to psychiatric disorders, cognitive or emotional disorders).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are older than 18 years of age diagnosed with acute mild ischemic stroke with large vessel occlusion (LVO-MIS) within 24 hours of onset will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Early neurological deterioration | 24 hours
  It is defined as an increase of ≥4 points from baseline NIHSS at hospital arrival, and excluding non-ischemic causes such as hemorrhagic transformation and epilepsy.

SECONDARY OUTCOMES:
Neurological functional outcome | 90 days
  Modified Rankin Scale (mRS) score is used to measure the degree of disability in patients who have had a stroke, as follows 0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Composite Temporal and spatial dynamic changes of the neurometabolites | acute stage (within 24 hours), the subacute stage (5-7 days) and the chronic stage (90 days)
  Signals of NAA, lactate, choline, creatine, and myo-inositol were evaluated using MRSI technology
Composite Temporal and spatial dynamic changes of the neurotransmitters | acute stage (within 24 hours), the subacute stage (5-7 days) and the chronic stage (90 days)
  Signal of GABA, glutamate, and glutamine determined by MRSI technology
Changes in whole-brain metabolic network connectivity | acute stage (within 24 hours), the subacute stage (5-7 days) and the chronic stage (90 days)
  Changes of metabolic connectivity mapping in whole brain between acute stage and chronic stage of stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Li Cao, phD, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No